CLINICAL TRIAL: NCT05105230
Title: Soluble Programmed Death 1 (sPD1) is a Diagnostic Biomarker of ILD in Patients With Rheumatoid Arthritis Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salwa Omar Mohammed, Resident doctor in Rhematology and rehabilitation department, Assiut University
Other Study IDs: sPD1 in RA
Record Dates: First submitted 2021-10-07; First posted 2021-11-03 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Interstitial lung disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: soluble programmed death 1biomarker — soluble programmed death 1biomarker

SUMMARY:
1. Evaluate the levels of serum (sPD1) in RA patients with ILD and those without.
2. Detect subclinical RA-ILD for early diagnosis and management of this devastating manifestation of RA

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic autoimmune disease that is characterized by a systemic inflammatory state that affects joints and other organs .

There are many types of RA-related pulmonary diseases. RA-related pulmonary diseases include airway disease such as bronchiolitis. There are interstitial lung diseases that include non-specific interstitial pneumonitis and usual interstitial pneumonia .

The pathogenesis of RA is multifactorial with contributions from genetic and environmental factors. (CD4+) T-cells is responsible for pro-inflammatory cytokines production and subsequent joint destruction .

The aetiology of RA-ILD may be related to smoking and other factors that activate autoimmunity and the attack of post-transcriptionally modified self-proteins, such as citrullinated peptides. Citrullinated peptide can be produced in the lungs of some patients, causing a pulmonary fibrosis .

Major subtypes of RA-ILD are defined by their histopathological or (HRCT) patterns

. Programmed death-1 belongs to CD28/B7 family and is expressed on the surface of activated T cells, B cells, NK cells, dendritic cells and Treg cells. sPD-1 is the soluble form of PD-1 that is obtained by phosphoric acid hydrolysis of membrane type PD-1 .

Programmed death-1 and its ligands are important negative regulators of the immune system. .

In RA, Persistent synovial T cell activation and inflammation may be reasoned to positive regulators overexpression, aberrant expression of negative regulators or functional antagonism of these molecules by soluble factors .

sPD-1 inhibits the PD-1/PD-L signalling pathway by interacting with PD-Ls and promotes the T cell activation .

ELIGIBILITY:
Inclusion Criteria:

* Adult RA Patients who fulfilled the 2010 ACR/European league against rheumatism (EULAR) criteria for the classification of RA (7).
* Adult RA patients with ILD (Nonspecific idiopathic interstitial pneumonia more than 16 years old).

Exclusion Criteria:

* Patients with other autoimmune diseases (systemic lupus erythematosus, polyarteritis nodosa sarcoidosis, dermatomyositis, scleroderma, spondylarthritis and inflammatory bowel disease).
* RA patients with lung affection other than ILD
* Patients with malignant tumors
* Patients with active infection
* Patients with severe heart, lung, and kidney dysfunction
* Patients with tuberculosis, pulmonary infection, chronic obstructive pulmonary disease, bronchiectasis, lung tumor, and pneumoconiosis disease.
* Uses of drugs (other than RA medication) known to cause ILD such as antimicrobial agents (Sulphonamide), cardiovascular agents (amiodarone) and Bromocriptine.

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1. Adult RA Patients
  2. Adult RA patients with ILD
  3. Adult healthy control
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
measure the levels of serum (sPD1)by ELISA in RA patients | baseline
  Evaluate the levels of serum (sPD1) in RA patients and its correlation with ILD

SECONDARY OUTCOMES:
early diagnosis of ILD in patients with RA | baseline
  Detect subclinical RA-ILD for early diagnosis and management of this devastating manifestation

REFERENCES:
- See also: Soluble Programmed Death Molecule 1 (sPD-1) As Predictor of Interstitial Lung Disease in Rheumatoid Arthritis — https://doi.org/10.21203/rs.3.rs-587880/v1
- See also: The PD-1/PD-L pathway in rheumatic diseases — https://doi.org/10.1016/j.jfma.2020.04.004
- See also: Clinical significance of soluble programmed death-1(sPD-1) in rheumatoid arthritis patients: Relation to disease activity and functional status — http://dx.doi.org/10.1016/j.ejr.2014.12.002